CLINICAL TRIAL: NCT06861166
Title: Randomized Controlled Study of Geranium Wilfordii Combined With Androgen Deprivation in Neoadjuvant Therapy for Prostate Cancer
Brief Title: Clinical Study of Geranium Wilfordii Combined With Androgen Deprivation in Neoadjuvant Therapy of Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: baotai Liang (Other)
Responsible Party: Sponsor-Investigator, baotai Liang, resident doctor, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZDSYLL512-Y01
Record Dates: First submitted 2025-03-02; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Prostate CA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geranium wilfordii combined with androgen deprivation treatment group (Experimental): Geranium wilfordii 15g decoction (Geranium 15g, decocted by the decocting machine in the decocting room of the pharmacy Department of the hospital) was taken orally, 200mL/ time, once/day, for 3 months + continuous androgen deprivation treatment.After completion of treatment, radical prostatectomy was performed 3 weeks later (±7 days).
  Interventions: Drug: Androgen deprivation treatment; Procedure: radical prostatectomy
- Androgen deprivation treatment group (Sham Comparator): Continuous androgen deprivation therapy.After completion of treatment, radical prostatectomy was performed 3 weeks later (±7 days).
  Interventions: Drug: Geranium wilfordii combined with androgen deprivation treatment; Procedure: radical prostatectomy

INTERVENTIONS:
Drug: Geranium wilfordii combined with androgen deprivation treatment — Geranium wilfordii 15g decoction (Geranium 15g, decocted by the decocting machine in the decocting room of the pharmacy Department of the hospital) was taken orally, 200mL/ time, once/day, for 3 months + continuous androgen deprivation treatment
  Arms: Androgen deprivation treatment group
Drug: Androgen deprivation treatment — Continuous androgen deprivation therapy
  Arms: Geranium wilfordii combined with androgen deprivation treatment group
Procedure: radical prostatectomy — After completion of treatment, radical prostatectomy was performed 3 weeks later (±7 days).

SUMMARY:
The high incidence of prostate cancer is one of the important diseases that threaten the health of old men in our country. Although androgen deprivation therapy is an important treatment option for prostate cancer, although neoadjuvant androgen deprivation therapy combined with radical prostatectomy reduced the positive rate of surgical margins, it did not show statistically significant improvement in prostate-specific antigen (PSA). At the same time, few trials reported pathological complete response (pCR) and minimal residual lesion (MRD).

The purpose of this project is to verify the efficacy of geranium combined with androgen deprivation in the treatment of locally advanced prostate cancer or oligometastatic prostate cancer before radical prostatectomy through randomized controlled clinical trials, so as to find an effective treatment for locally advanced prostate cancer or oligometastatic prostate cancer.

DETAILED DESCRIPTION:
This study will divide patients into two sections, and eligible patients will be enrolled. Patients with locally advanced prostate cancer or oligo-metastatic prostate cancer were divided into geranium combined androgen deprivation therapy group and androgen deprivation therapy group according to a computer-generated random sequence. In the treatment group, except for continuous androgen deprivation treatment, geranium geranium decoction was taken orally every day; The control group only received continuous androgen deprivation therapy, and the usage was the same as the treatment group. After starting the intervention, all patients should be followed up in our hospital 7, 14, 28, 56, 84 days after treatment to review blood PSA and other indicators. At the end of the treatment, imaging examinations were followed up and radical prostatectomy was performed 3 weeks later (±7 days).

ELIGIBILITY:
Inclusion Criteria:

* ① Age ≥18 years and ≤85 years;

  * Histologically confirmed prostate cancer without small cell features;

    * Metastatic prostate cancer was identified by imaging examination with ≤5 oligometastases (bone or lymph node metastases) or cT3-4 stages; ④The score of ECOG (Eastern Cooperative Oncology Group) was 0-1; ⑤ All patients voluntarily sign informed consent, and can adhere to treatment and follow-up;

Exclusion Criteria:

* ①Any previous or ongoing PCa treatment, including radiotherapy, chemotherapy, ADT, etc.

  * Previous prostatectomy;

    * Any other serious basic medical, mental, psychological, and other diseases that, in the judgment of the investigator, may affect the treatment of the patient

      * Allergic to the drugs used; ⑤ Refuse to undergo radical prostatectomy; ⑥ According to the investigator's judgment, it is not suitable to participate in this clinical trial;

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
pCR or MRD rate | up to 4 weeks
  pCR (pathological complete response) is defined as cancer that is not morphologically recognizable in a prostatectomy specimen; MRD (small residual lesion) was defined as the maximum cross-section size of the residual tumor ≤5 mm, and RCB (residual cancer load) ≤ 0.25cm3 (tumor volume ≤ 0.5cm3 × tumor cells ≤ 50%) was used to calculate the tumor volume through three-dimensional volume estimation according to the maximum cross-section size and number of cross-sections involved in the tumor. Correction of tumor cell structure;

SECONDARY OUTCOMES:
PSA level change | At the end of Cycle 1 and Cycle 2 (each cycle is 21 days)
Biochemical progression-free survival after radical prostatectomy | The evaluation period was up to 1 year ( from the date of completion of surgery to the date of first recorded psa progression)
Pathologic responses after radical prostatectomy (including positive surgical margin, tumor size, prostatic extension, seminal vesicle infiltration, and lymph node involvement) | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vice President of Zhongda Hospital, Study Director — Zhongda Hospital

IPD SHARING:
Plan to Share IPD: No